CLINICAL TRIAL: NCT07111689
Title: Virtual Reality for Cognitive Enhancement in Schizophrenia: A Randomized Controlled Trial
Brief Title: The Effect of Virtual Reality on Cognitive Skills in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Berkan Torpil, PhD, Assoc Prof, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/10
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Ability General; Virtual Reality; Virtual Reality Cognitive Training; Schizophrenia Disorder
Keywords: schizoprenia; virtual reality; cognitive
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): cognitive rehabilitation with conventional occupational therapy intervention
  Interventions: Behavioral: Conventional Occupational Therapy Interventiın
- Study Group (Experimental): virtual reality intervention in addition to conventional occupational therapy intervention
  Interventions: Behavioral: Conventional Occupational Therapy Interventiın; Behavioral: Virtual Reality İntervention

INTERVENTIONS:
Behavioral: Conventional Occupational Therapy Interventiın — 1-2. Week: Occupation-based interventions for visual skills 3-6. Week: Social Skills Training 7-8. Week: Interventions for participation problems in ADLs
Behavioral: Virtual Reality İntervention — In this study, the Xbox 360 gaming console and Kinect sensor were utilized for the virtual reality (VR) intervention. The Xbox 360 functions as an interactive gaming platform, while the Kinect sensor is a motion-detection device that captures users' positions and movements through an integrated camera and sensors. The selection of games for the VR intervention was conducted in collaboration with experts from various disciplines. The evaluation process considered the cognitive and functional demands required for successful gameplay, the potential skills each game could enhance, and the overall therapeutic purpose of the selected games. Following an independent assessment of each game, nine games were identified as suitable for the intervention. Given that all selected games shared similar functional requirements, participants were provided access to the full set of games to optimize engagement and motivation.
  Arms: Study Group

SUMMARY:
This study was conducted to examine the effect of virtual reality intervention, given in addition to conventional occupational therapy intervention, on general cognitive functions (attention, orientation, memory, visual skills, visual-motor skills, praxis, executive functions, etc.) in individuals with schizophrenia. This study was designed in accordance with the CONSORT statement, which standardizes randomized controlled trials. Additionally, the study was approved by a university's scientific research ethics committee.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled trial and conducted using the CONSORT checklist. Individuals who met the inclusion and exclusion criteria were included in the study. Both groups received traditional occupational therapy intervention, while the intervention group also received virtual reality intervention. All intervention procedures in the study were planned to take place three days a week for eight weeks, with each session lasting 45 minutes. A total of 114 individuals were included in the study; 54 were in the control group and 60 were in the intervention group.

Interventions

Conventional occupational therapy intervention approach was applied in both groups. The intervention group additionally received VR application with Microsoft Xbox 360 and Kinect. The interventions consisted of 45-minute sessions 3 days a week for 8 weeks. The intervention procedures are described in detail below and all interventions were performed by the last author of the study :

Conventional Occupational Therapy Intervention:

1-2. Week: Occupation-based interventions for visual skills Within the framework of the occupational therapy intervention calendar, in the first two weeks, participants were given training on visual memory, figure-ground perception, visual discrimination, visual completion, spatial perception, etc., which are the sub-parameters of visual perception skills. It is aimed to increase the visual skill levels of people by making interventions to improve the parameters. Response plan; As a result of the participants' occupation preferences and evaluation results, it was created and implemented using client-centered occupations that aim to increase people's visual skill levels.

3-6. Week: Social Skills Training In these weeks, it was aimed to develop different social skill levels of the participants by using various occupations related to the problematic areas of social skills with personalized targeted occupations. Within the framework of the intervention plan, various activities were prepared to develop skills such as "listening to others, making requests, expressing positive emotions and expressing unpleasant emotions", which are among the basic social skills areas. In addition, social skills parameters such as communication skills, assertiveness skills, conflict management skills, social life skills, friendship skills, interpersonal skills, health maintenance skills, professional/work skills were also included in the intervention plan. During these weeks, social skills were practiced with different tasks and sequential operations, and the development of memory, attention, orientation, praxis and executive skills was also aimed.

7-8. Week: Interventions for participation problems in ADLs Participants' problems in ADLs were identified through client-centered interviews and assessments, and their participation problems were evaluated in terms of personal, environmental and occupation-related factors. It was aimed to solve these problems by applying a holistic client-centered intervention approach to participation problems. During these weeks, the client-centered intervention approach aimed to improve cognitive functions, especially at the level of executive skills such as problem solving, time management, task initiation and completion.

VR Intervention Procedure In this study, the Xbox 360 gaming console and Kinect sensor were utilized for the virtual reality (VR) intervention. The Xbox 360 functions as an interactive gaming platform, while the Kinect sensor is a motion-detection device that captures users' positions and movements through an integrated camera and sensors.

The selection of games for the VR intervention was conducted in collaboration with experts from various disciplines. The evaluation process considered the cognitive and functional demands required for successful gameplay, the potential skills each game could enhance, and the overall therapeutic purpose of the selected games. Following an independent assessment of each game, nine games were identified as suitable for the intervention. Given that all selected games shared similar functional requirements, participants were provided access to the full set of games to optimize engagement and motivation. The specific games and the cognitive functions they target are detailed in Appendix 1.

The intervention was conducted in a designated unit with a total area of approximately 30 m². To mitigate the risk of falls, the flooring of the intervention space was covered with a soft, impact-absorbing surface.

ELIGIBILITY:
Inclusion Criteria:

* (1) age between 18 and 65 years,
* (2) Participants must have been diagnosed with Schizophrenia according to the ICD-10 diagnostic criteria,
* (3) Participants must be able to read and write at a level that will allow them to understand the content of the study,
* (4) There must be no severe cognitive impairment diagnosed that would prevent participation in the study,
* (5) Participants' antipsychotic treatments must be stable (no medication changes in the last 3 months),
* (6) Participants must be competent to provide informed consent

Exclusion Criteria:

* (1) Existence of additional diagnoses such as schizoaffective disorder, bipolar disorder or severe depressive disorder,
* (2) Existence of active substance or alcohol addiction diagnosed in the last 6 months,
* (3) Presence of diseases that may affect cognitive functions such as epilepsy, dementia, Parkinson's disease,
* (4) Exclusion of individuals who have active psychotic episodes or severe agitation during the study period,
* (5) Exclusion of individuals who are at risk of harming themselves or others,
* (6) For female participants, there is pregnancy or breastfeeding,
* (7) There are conditions such as visual or hearing impairment that may prevent active participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-21 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
The Loewenstein Occupational Therapy Cognitive Assessment (LOTCA) | 1 hour
  The LOTCA is a performance test that consists of 20 items. The test includes testing materials such as card decks, colored blocks, a pegboard set, and other items. Additionally, a manual is provided that defines the cognitive domains assessed and provides administration instructions, and specific scoring guidelines. The LOTCA was scored on a Likert-type scale from 1 to 4, except for items 1-5 which related to categorization, unstructured Risk Object Classification, and structured Risk Object Classification. Higher scores indicate better cognitive functions

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Science, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No